CLINICAL TRIAL: NCT03449550
Title: Validity and Cost-effectiveness Analysis of a Home Respiratory Polygraphy for the Diagnosis of Obstructive Sleep Apnea in Children (DINISAS)
Brief Title: Validity of a Home Respiratory Polygraphy for the Diagnosis of Obstructive Sleep Apnea in Children (DINISAS)
Acronym: DINISAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); ResMed (Industry); Complejo Hospitalario de Caceres (Other); Hospital Universitario de Burgos (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital de Basurto (Other); Hospital Vall d'Hebron (Other); Fundación Jimenez Diaz de Madrid (Unknown); Hospital Universitario La Paz (Other); Hospital Universitario 12 de Octubre (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital de Guadalajara (Unknown); University of Chicago (Other)
Responsible Party: Principal Investigator, Joaquin Duran-Cantolla, MD, Principal Investigator. MD,PhD, Hospital Universitario Araba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI14/01187
Record Dates: First submitted 2017-10-06; First posted 2018-02-28 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Child obstructive sleep apnea; Home Respiratory Polygraphy; Diagnosis; Validity; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disease | interventions — Reproducibility of Results

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnostic Randomizing (Active Comparator): Randomizing to start with home respiratory polygraphy (HRP) or Standard Polysomnography (PSG)
  Interventions: Other: Home Respiratory Polygraphy (HRP); Other: Standard Polysomnography (PSG)
- Therapeutic Randomizing (Active Comparator): Randomizing for therapeutic decision taken with home respiratory polygraphy (HRP) or Standard Polysomnography (PSG)
  Interventions: Other: Home Respiratory Polygraphy (HRP); Other: Standard Polysomnography (PSG)

INTERVENTIONS:
Other: Home Respiratory Polygraphy (HRP) — Randomizing to start with home respiratory polygraphy
  Other Names: Validity
  Arms: Diagnostic Randomizing
Other: Standard Polysomnography (PSG) — Randomizing to start with Standard Polysomnography (PSG)
  Other Names: Validity
  Arms: Diagnostic Randomizing
Other: Home Respiratory Polygraphy (HRP) — Randomizing for therapeutic decision taken with home respiratory polygraphy (HRP)
  Other Names: Effectiveness
  Arms: Therapeutic Randomizing
Other: Standard Polysomnography (PSG) — Randomizing for therapeutic decision taken with Standard Polysomnography (PSG)
  Other Names: Effectiveness
  Arms: Therapeutic Randomizing

SUMMARY:
To assess the diagnostic validity and cost-effectiveness of a home respiratory polygraphy (HRP) performed at home compared with the standard polysomnography (PSG) in children with clinically suspected Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
AIMS: To assess the diagnostic validity and cost-effectiveness of a home respiratory polygraphy (HRP) performed at home compared with the standard polysomnography (PSG) in children with clinically suspected Obstructive Sleep Apnea (OSA).

METHODOLOGY: DESIGN: Randomized, prospective, multicenter, double blind and crossover trial. The study will include 320 children, both sexes, with clinical suspicion of obstructive sleep apnea (OSA). MEASUREMENTS: To all patients with clinical suspected OSA and referred to the sleep units, the following questionnaires and measurements will be performed: a) clinic history; b) Anthropometric variables: weight, height, body mass index, neck circumference and percentile; c) Chervin questionnaire, quality of life and clinical questionnaires and comorbidity; d) PSG in the sleep laboratory; e) HRP at home; f) Quantitative unbiased proteinic urine analysis and g) Cost-effectiveness variables.

ANALYSIS: Data from HRP and from full PSG will be compared as follows: 1) Agreement of results according to the different apnea-hypopnea index by using the ROC curves; 2) The concordance of the diagnosis and treatment decisions when using clinical findings and data from PSG or HRP at home, 3) All data will be analyzed independently by participating hospitals according the Cohen Kappa method, 4) A diagnosis paradigm based on proteinic defined variables and 5) A cost-effectiveness analysis of the different diagnostic and therapeutic procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 14 years of age of both sexes consecutively assessed for clinical suspicion of OSA, defined as: snoring children with observed respiratory and / or apnea pauses and / or ventilatory effort during observed sleep, and who were asked for a sleep test
* Written informed consent signed.

Exclusion Criteria:

* Place of residence more than 100 km from the hospital
* Psychophysical incapacity to perform the study at home
* Severe, unstable or exacerbated cardio-vascular, cerebro-vascular or respiratory disease, that makes it impossible to carry out adequate studies
* Children with chronic insomnia and / or depressive syndrome
* Children with malformative syndromes, Down Syndrome and neuromuscular diseases
* Complete or near complete nasal obstruction that prevents obtaining a quality signal with the HRP
* History of surgery and / or previous Positive continuous pressure (CPAP) for OSA

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic validity of a Home Respiratory Polygraphy (HRP) | baseline
  To establish the diagnostic validity of home respiratory polygraphy (HRP) compared with the findings obtained with polysomnography (PSG) in the sleep laboratory in children with suspected Obstructive Sleep Apnea (OSA), based on the results of Apnea-hypopnea Index (AHI)

SECONDARY OUTCOMES:
Cost effectiveness analysis | baseline
  Cost-efficacy evaluation: the analysis will be made in both arms based on intention to treat. Only direct costs will be analyzed: the cost of the use of polysomnography and home respiratory polygraphy (Staff and consumable material).
Validation of the therapeutic decision | 6 month
  Analyze the concordance in the therapeutic decision using clinical findings and the results of Apnea-Hypopnea Index (AHI) from standard polysomnography (PSG) compared with data from home respiratory polygraphy (HRP)
Validity of the determination of a protein sequence in urine in OSA | baseline
  To analyze the validity of the determination of a protein sequence in urine, alone or in combination, to establish the diagnosis of OSA and to evaluate its modification over time after the treatment of OSA
Pediatric Sleep Questionnaire. | baseline and at six month
  Pediatric Sleep Questionnaire designed to screen for sleep problems in children.The scale consists of 22 parent-reported items examining snoring and breathing problems, daytime sleepiness, inattention, hyperactivity, and other signs and symptoms of apnea including obesity and nocturnal enuresis.
  The result is a number, a proportion that ranges from 0.0 to 1.0. Scores >0.33 are considered positive and suggestive of high risk for a pediatric sleep-related breathing disorder
BEARS Sleep screening | baseline and at six month
  BEARS Sleep screening is divided into five major sleep domains (B=Bedtime Issues, E=Excessive Daytime Sleepiness, A=Night Awakenings, R=Regularity and Duration of Sleep, S=Snoring), providing a comprehensive screen for the major sleep disorders affecting children in the 2- to 18-year old range
Quality of life (KINDLR) | baseline and at six month
  The KINDLR is a generic instrument for assessing Health-Related Quality of Life in children and adolescents aged 3 years and older. Consists of 24 Likert-scaled items associated with six dimensions: physical well-being, emotional well-being, self-esteem, family, friends and everyday functioning (school). The response categories cover 3 levels (1=never, 2=sometimes, 3=very often)
Children's sleep habits questionnaire (CSHQ) | baseline and at six month
  Parent-report sleep screening instrument designed for school-aged children.The instrument evaluates the child's sleep based on behavior within eight different subscales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness.
Anthropometric variables | baseline and at six month
  Body mass index
Blood pressure | baseline and at six month
  Blood pressure measurements: systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Alava, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luz Alonso-Alvarez M, Canet T, Cubell-Alarco M, Estivill E, Fernandez-Julian E, Gozal D, Jurado-Luque MJ, Lluch-Rosello MA, Martinez-Perez F, Merino-Andreu M, Pin-Arboledas G, Roure N, Sanmarti FX, Sans-Capdevila O, Segarra-Isern F, Tomas-Vila M, Teran-Santos J; Sociedad Espanola de Sueno; Area de Sueno de la Sociedad Espanola de Neumologia y Cirugia Toracica(SEPAR)]. [Consensus document on sleep apnea-hypopnea syndrome in children (full version). Sociedad Espanola de Sueno. El Area de Sueno de la Sociedad Espanola de Neumologia y Cirugia Toracica(SEPAR)]. Arch Bronconeumol. 2011 May;47 Suppl 5:0, 2-18. doi: 10.1016/S0300-2896(11)70026-6. Epub 2011 Jun 22. No abstract available. Spanish. PMID 22682520
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J et al. American Academy of Pediatrics Statement. Clinical practice guideline: diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics109:704-23, 2002.
- [Background] Alonso-Alvarez ML, Cordero-Guevara JA, Teran-Santos J, Gonzalez-Martinez M, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Kheirandish-Gozal L, Gozal D. Obstructive sleep apnea in obese community-dwelling children: the NANOS study. Sleep. 2014 May 1;37(5):943-9. doi: 10.5665/sleep.3666. PMID 24790273
- [Background] Gileles-Hillel A, Alonso-Alvarez ML, Kheirandish-Gozal L, Peris E, Cordero-Guevara JA, Teran-Santos J, Martinez MG, Jurado-Luque MJ, Corral-Penafiel J, Duran-Cantolla J, Gozal D. Inflammatory markers and obstructive sleep apnea in obese children: the NANOS study. Mediators Inflamm. 2014;2014:605280. doi: 10.1155/2014/605280. Epub 2014 Jun 1. PMID 24991089
- [Background] Reuveni H, Simon T, Tal A, Elhayany A, Tarasiuk A. Health care services utilization in children with obstructive sleep apnea syndrome. Pediatrics. 2002 Jul;110(1 Pt 1):68-72. doi: 10.1542/peds.110.1.68. PMID 12093948
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Spruyt K, Gozal D. Screening of pediatric sleep-disordered breathing: a proposed unbiased discriminative set of questions using clinical severity scales. Chest. 2012 Dec;142(6):1508-1515. doi: 10.1378/chest.11-3164. PMID 22677350
- [Background] Nixon GM, Kermack AS, Davis GM, Manoukian JJ, Brown KA, Brouillette RT. Planning adenotonsillectomy in children with obstructive sleep apnea: the role of overnight oximetry. Pediatrics. 2004 Jan;113(1 Pt 1):e19-25. doi: 10.1542/peds.113.1.e19. PMID 14702490
- [Background] Marcus CL, Keens TG, Ward SL. Comparison of nap and overnight polysomnography in children. Pediatr Pulmonol. 1992 May;13(1):16-21. doi: 10.1002/ppul.1950130106. PMID 1589307
- [Background] Goodwin JL, Enright PL, Kaemingk KL, Rosen GM, Morgan WJ, Fregosi RF, Quan SF. Feasibility of using unattended polysomnography in children for research--report of the Tucson Children's Assessment of Sleep Apnea study (TuCASA). Sleep. 2001 Dec 15;24(8):937-44. doi: 10.1093/sleep/24.8.937. PMID 11766164
- [Background] Jacob SV, Morielli A, Mograss MA, Ducharme FM, Schloss MD, Brouillette RT. Home testing for pediatric obstructive sleep apnea syndrome secondary to adenotonsillar hypertrophy. Pediatr Pulmonol. 1995 Oct;20(4):241-52. doi: 10.1002/ppul.1950200407. PMID 8606854
- [Background] Moss D, Urschitz MS, von Bodman A, Eitner S, Noehren A, Urschitz-Duprat PM, Schlaud M, Poets CF. Reference values for nocturnal home polysomnography in primary schoolchildren. Pediatr Res. 2005 Nov;58(5):958-65. doi: 10.1203/01.PDR.0000181372.34213.13. Epub 2005 Sep 23. PMID 16183829
- [Background] Alonso Alvarez ML, Teran Santos J, Cordero Guevara JA, Navazo Eguia AI, Ordax Carbajo E, Masa Jimenez JF, Pelayo R. [Reliability of respiratory polygraphy for the diagnosis of sleep apnea-hypopnea syndrome in children]. Arch Bronconeumol. 2008 Jun;44(6):318-23. Spanish. PMID 18559221
- [Background] Brockmann PE, Schaefer C, Poets A, Poets CF, Urschitz MS. Diagnosis of obstructive sleep apnea in children: a systematic review. Sleep Med Rev. 2013 Oct;17(5):331-40. doi: 10.1016/j.smrv.2012.08.004. Epub 2013 Jan 30. PMID 23375659
- [Background] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- [Background] Tan HL, Gozal D, Kheirandish-Gozal L. Obstructive sleep apnea in children: a critical update. Nat Sci Sleep. 2013 Sep 25;5:109-23. doi: 10.2147/NSS.S51907. PMID 24109201
- [Background] Ragette R, Wang Y, Weinreich G, Teschler H. Diagnostic performance of single airflow channel recording (ApneaLink) in home diagnosis of sleep apnea. Sleep Breath. 2010 Jun;14(2):109-14. doi: 10.1007/s11325-009-0290-2. Epub 2009 Aug 28. PMID 19714380
- [Background] Masa JF, Duran-Cantolla J, Capote F, Cabello M, Abad J, Garcia-Rio F, Ferrer A, Mayos M, Gonzalez-Mangado N, de la Pena M, Aizpuru F, Barbe F, Montserrat JM; Spanish Sleep Network; Larrateguy LD, de Castro JR, Garcia-Ledesma E, Utrabo I, Corral J, Martinez-Null C, Egea C, Cancelo L, Garcia-Diaz E, Carmona-Bernal C, Sanchez-Armengol A, Fortuna AM, Miralda RM, Troncoso MF, Monica G, Martinez-Martinez M, Cantalejo O, Pierola J, Vigil L, Embid C, Del Mar Centelles M, Prieto TR, Rojo B, Vanesa L. Effectiveness of home single-channel nasal pressure for sleep apnea diagnosis. Sleep. 2014 Dec 1;37(12):1953-61. doi: 10.5665/sleep.4248. PMID 25325484
- [Background] Gozal D, Jortani S, Snow AB, Kheirandish-Gozal L, Bhattacharjee R, Kim J, Capdevila OS. Two-dimensional differential in-gel electrophoresis proteomic approaches reveal urine candidate biomarkers in pediatric obstructive sleep apnea. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1253-61. doi: 10.1164/rccm.200905-0765OC. Epub 2009 Sep 24. PMID 19797158